CLINICAL TRIAL: NCT06413914
Title: Evaluation of Cognitive Behavioral Therapy for Long-term Pain in Rheumatic Disease, Including Validation the Questionnaire of AE-FS
Brief Title: Evaluation of Cognitive Behavioral Therapy for Long-term Pain in Rheumatic Disease, Including Validation of AE-FS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Kåre Osnes, Researcher PhD MD, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS-00805; 656858 (Registry Identifier: REK)
Record Dates: First submitted 2024-01-17; First posted 2024-05-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Rheumatic Diseases; Pain, Chronic
Keywords: "Cognitive behavioral therapy"; Long-term pain; Avoidance-Endurance Questionnaire; Rheumatic disease
MeSH Terms: conditions — Rheumatic Diseases; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: 200 patients with long-term pain and rheumtic disease, participate in cognitive behavioral therapy individually or in a group. The treatment consists of 8 sessions, 7 weekly sessions and a booster session 2 months after the end of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive behavioral Therapy (Experimental): Cognitive behavioral therapy is the psychological approach in this study. It is associated with better outcomes of rehabilitation for long-term pain in general, reduced pain intensity and less use of medication and health services, sustaining factors that provide an understanding of how thoughts and feelings affect the experience of pain. An important aim is also a reduction in pain-related rumination and worry and changed metacognition that maintains inhibiting behavior and thought patterns.
  A workbook for pain has been developed. It contains knowledge about pain and pain management, describes measures and homework from session to session. The treatment consists of 8 sessions with 7 weekly sessions + 1 booster session 2 months after the end of treatment.
  Interventions: Behavioral: Cognitive behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral Therapy — Cognitive behavioral therapy is the psychological approach in this study. It is associated with better outcomes of rehabilitation for long-term pain in general, reduced pain intensity and less use of medication and health services, sustaining factors that provide an understanding of how thoughts and feelings affect the experience of pain. An important aim is also a reduction in pain-related rumination and worry and changed metacognition that maintains inhibiting behavior and thought patterns.
  A workbook for pain has been developed. It contains knowledge about pain and pain management, describes measures and homework from session to session. The treatment consists of 8 sessions with 7 weekly sessions + 1 booster session 2 months after the end of treatment.
  .

SUMMARY:
Catastrophic thinking is a risk factor for a poor prognosis for pain in general and rheumatic disease in particular, which for many contributes to a behavioral pattern characterized by avoidance. Other people with long-term pain, on the other hand, have a pattern where they suppress thoughts and feelings of fear associated with pain, and push themselves to carry out activities. An inappropriate form of endurance can help maintain and intensify pain. The AE-FS is a short version of the Avoidance-Endurance Questionnaire with different subscales for maintaining activity despite pain. AE-FS can be of great clinical utility. The study of patients with rheumatic disease and long-term pain will validate a Norwegian version of the AE-FS as well as examine how the AE-FS seen in connection with other relevant questionnaires, including the Pain Catastrophizing Scale , reflects mechanisms for change in cognitive behavioral therapy for long-term pain. The effect of the intervention is evaluated with questionnaires at baseline/start of treatment, end of treatment, two months after end of treatment and after six months.

DETAILED DESCRIPTION:
Background for the project Up to 30% of the adult population in Norway state that they have had long-term pain . Long-term pain in the musculoskeletal system accounts for 50% of disability cases and is the most frequent cause of long-term absence. This group includes rheumatic disease, back and neck disorders, pelvic pain and shoulder problems. Rheumatic disease is a collective term for over 200 different diseases that are divided into inflammatory rheumatic disease (arthritis, spondyloarthritis, psoriatic arthritis, connective tissue diseases and vasculitis), degenerative diseases (arthrosis) and soft tissue rheumatism (fibromyalgia). Fibromyalgia is characterized by widespread and long-lasting muscle pain and occurs in about 5% of the population.

The pain picture in rheumatic disease is complex with different pain mechanisms and frequent comorbidity with sleep difficulties, fatigue and psychological problems. The pain can be linked to inflammation and to structural changes, but also to changes in the central nervous system.

With support from Stiftelsen Dam, the Unit for mental health services in somatics and the Unit for research and innovation at the Adult Psychiatric Department Vinderen and the Clinic for Rheumatology, Outpatient Clinic and Research, Diakonhjemmet Hospital, have developed an intervention based on clinical health psychology and cognitive behavioral therapy. The target group is primarily patients with long-term pain and rheumatic disease. The treatment is described in a chapter in the Handbook of Clinical Health Psychology .

A workbook for pain has been developed, following revisions and feedback from 15 individual patients and participants in 2 treatment groups (one physical and one digital) who have followed the scheme. The workbook contains knowledge about pain and pain management, describes measures and homework from session to session. The treatment offered in the project spans 8 sessions of 2 hours each and is carried out either digitally or by physical attendance. A corresponding manual has also been developed for individual treatment over approx. 10 sessions of 45 minutes. The patients are called in for a follow-up appointment 2 months after the ordinary termination.

Negative thought and reaction and behavior patterns in long-term pain Catastrophic thinking is an inappropriate coping style where one overestimates the threat of pain, ponders the causes and is worried about the consequences. In arthritis, catastrophic thinking predicts more intense pain and severe depression symptoms and poorer physical function . In knee osteoarthritis, catastrophizing predicts a longer postoperative course in hospital, and more avoidance of physical activity .

Some patients suppress thoughts associated with pain or the fear of it and push themselves to carry out activities. It represents an inappropriate and inflexible form of endurance, which can contribute to maintaining and intensifying pain.

The short version AE-FS can be of great clinical value. A patient with high scores on the questionnaire may be in a vicious circle which in the long term increases pain and affects quality of life. The patient ignores the pain or the fear of it, and does not pay necessary attention to it. The form consists of 9 statements, 7 of them on two scales for mild and severe pain, respectively, where you must indicate whether and how often you have acted in this way in the last two weeks. Examples of statements are:

"When I am in pain

* I try not to take any notice of it.
* I clench my teeth.
* keep appointments even though I don't feel up to it.

There are 7 answer options (never, almost never, seldom, sometimes, often, mostly and always). In addition, the patients are asked to indicate their mood and the possibility of depressive symptoms in the last two weeks, more specifically if they enjoy things just as ever and think they make decisions about as well as ever.

Issues for the study

1. The AE-FS questionnaire can be of great clinical value for mapping behavior and thoughts in mild and severe pain, both to predict long-term pain and as an educational tool in the treatment of patients. In the project, we will validate the form, by assessing its suitability for our patient group and compliance with other validated forms which, among other things, measure pain, depressive symptoms, anxiety symptoms and function.
2. In the project, we also want to evaluate the feasibility and effect of the treatment for:

   1. Pain, measured by the Brief Pain Inventory questionnaire - short form (Cleeland & Ryan, 1994)
   2. General symptoms, measured by the PROMIS-29 questionnaire (Patient reported outcomes measurement information system).
   3. Quality of life/general health, measured by the EQ-5D-5L questionnaire (general health questionnaire).
   4. Any other relevant questionnaires.
   5. Feasibility and satisfaction, including attendance, dropouts, etc.
3. We also want to investigate whether negative thought and reaction and behavior patterns in long-term pain measured by AE-FS and/or PCS can predict and/or mediate treatment response when it comes to pain.
4. We also want to evaluate other possible predictors of treatment response, such as age, sex, duration of pain, etc.

Method and implementation In the study, we will evaluate the effect of the intervention using questionnaires at baseline, at the start of treatment, at the end of treatment, at the booster time two months after the end of treatment and 6 months later.

Suitable forms have been assessed in consultation with the reference group. We use the following forms:

Brief Pain Inventory - short form ; PROMIS-29 (Patient reported outcomes measurement information system); generic EQ-5D-5L (general health and quality of life questionnaire), PCS (Pain Catastrophizing Scale), AE-FS (The avoidance-endurance questionnaire - short form, ), and four questions from the MCQ (MetaCognition Questionnaire) about positive assumptions about worry and an assumption that worry cannot be controlled, respectively. Patients must also fill in a background form upon inclusion with, among other things, demographic variables, and possibly simple "anchor questions" aimed directly at current issues.

We will also register attendance and non-attendance, possibly from the patient record.

Treatment within the project Cognitive behavioral therapy is the psychological approach that has the best evidence for long-term pain in general, and which is highlighted as a theoretical framework in EULAR's recommendations for patient education in rheumatic disease.

Cognitive behavioral therapy is associated with better outcomes of rehabilitation for long-term pain in general, reduced pain intensity and less use of medication and health services.

There is evidence that exposure therapy aimed at pain-related avoidance behavior reduces the symptoms of fibromyalgia . Work with pain-related imagery as well as motivation, goals and values and measures to strengthen compliance when using rules of action are also included. In addition, measures are taken to influence patterns of action characterized by inappropriate endurance and accompanying overload.

Participants in the study/preparedness throughout the project period We plan to include up to 200 patients who participate in the treatment plan, either individually or treated in a course/group at the Unit for mental health services in somatics, Diakonhjemmet hospital. The patients included have both a rheumatic disorder and a long-term pain condition.

All patients have an assessment interview with a psychologist associated with the project, before starting the treatment. There they will receive information about the treatment and the research project. They are told that participation in the project is voluntary and that it is perfectly fine to receive the treatment without participating in the research. If they then express that they are interested in participating in the research project, they will receive written and verbal information about the project (consent form), and information that, prior to the start of treatment, they will receive a link via SMS, where they can sign the consent and fill in the questionnaires. Alternatively, in the assessment interview, they will be given a written consent form and the questionnaires which they can hand in to the researchers in the study, possibly sending in a pre-stamped envelope.

The included questionnaires are completed at inclusion/start of treatment, end of treatment, at the follow-up appointment 2 months after the end of ordinary treatment and 6 months later. In order to ensure privacy and good quality of the answers, the research participants are informed that the forms should be completed in quiet surroundings without public exposure. In the consent form, they will also receive information that the forms will only be used in the research and that they can contact the project manager throughout the project period if filling in the forms would result in negative reactions or the need for clarifying conversations. If necessary, they can have a conversation with the psychologist responsible for the treatment.

Project group The project group for the study is divided into two parts, where the psychologists Elin Fjerstad, Torkil Berge and Ingrid Hyldmo are responsible for the development and implementation of the treatment and the researchers Kåre Osnes (project manager), Selle Aarrestad Provan, Rikke Helene Moe, Bente Bull-Hansen and Andrew Malcolm Garratt are responsible for the research part of the project. Everyone in the research group is employed at Diakonhjemmet hospital.

Handling of data Patients fill in the questionnaires digitally via Nettskjema/TSD, alternatively on paper.

The data that is collected on paper is stored de-identified and locked in the office of the project employee/archive. The data is transferred de-identified and stored on an access-controlled research server. The code list is stored in a separate access-controlled folder on the research server, where only the project manager and employees responsible for research logistics have access. The data will be anonymised (the code list will be deleted and other personally identifiable information will be removed) no later than five years after the end of the project (the end of the project is tentatively 31 December 2030).

The data that is collected digitally via Nettskjema/TSD is transferred to an access-controlled folder in the research server.

According to the new General Data Protection Regulation (GDPR), the controller at Diakonhjemmet hospital and project manager Kåre Osnes has an independent responsibility to ensure that the processing of personal data has legal basis. This project has legal basis in the EU's GDPR article 6 no. 1a and article 9 no. 2a, consent. The project will be assessed by the data protection representative and the research committee at Diakonhjemmet hospital.

The results will be published in scientific journals, through the user organisations' magazines and websites, and spread through social media.

The project is a collaborative project between the Department of Adult Psychiatry and the Center for treatment of Rheumatic and Musculoskeletal Diseases (REMEDY).

REMEDY is an interdisciplinary research center led by Diakonhjemmet hospital in partnership with Oslo University Hospital. The research center aims to improve the treatment of musculoskeletal diseases and has a particular focus on intervention studies in people with auto-immune rheumatic diseases. The center is funded by the Research Council, which is a research center for clinical treatment, and by the Olav Thon Foundation

Schedule

Course and processing with collection of personal data: 2024-2027 Analyzes of research data: 2027-2028 Publication with writing of articles 2028-2030

ELIGIBILITY:
Inclusion Criteria:

* A rheumatic disorder and a long term pain condition
* Written consent

Exclusion Criteria:

* Participation in another therapy during the study periode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of AE-FS | 8 months
  1. The AE-FS questionnaire can be of great clinical value for mapping behavior and thoughts in mild and severe pain, both to predict long-term pain and as an educational tool in the treatment of patients. In the project, we will validate the form, by assessing its suitability for our patient group and compliance with other validated forms which, among other things, measure pain, depressive symptoms, anxiety symptoms and function.
Evaluation of cognitive behavioral therapy for long-term pain in rheumatic disease - Feasibility | 8 months
  In the project, we also to evaluate the feasibility of the treatment:Feasibility and satisfaction, including attendance, dropouts, etc.
Evaluation of cognitive behavioral therapy for long-term pain in rheumatic disease - Pain | 8 months
  Pain, measured by the Brief Pain Inventory questionnaire - short form
Evaluation of cognitive behavioral therapy for long-term pain in rheumatic disease - General symptoms | 8 months
  General symptoms, measured by the PROMIS-29 questionnaire (Patient reported outcomes measurement information system).
Evaluation of cognitive behavioral therapy for long-term pain in rheumatic disease - Quality of life | 8 months
  Quality of life/general health, measured by the EQ-5D-5L questionnaire (general health questionnaire).

SECONDARY OUTCOMES:
Analyses of predictors and mediators | 8 months
  3. We also want to investigate whether negative thought and reaction and behavior patterns in long-term pain measured by AE-FS and/or PCS can predict and/or mediate treatment response when it comes to pain.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Soegaard, PhD, Study Chair — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Sykehus, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researshers